CLINICAL TRIAL: NCT07171450
Title: Computerized Cognitive Remediation of Postviral Neurocognitive Dysfunction in Older Adults
Brief Title: Cognitive Remediation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cutter Lindbergh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Cutter Lindbergh, Assistant Professor, UConn Health
Organization: UConn Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-389-2; 1K23AG086612-01A1 (NIH)
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Aging; Inflammation; Cognitive Remediation; Cognitive Dysfunction; Postviral Syndrome; Digital Medicine
Keywords: Aging; Inflammation; Cognitive Remediation; Cognitive dysfunction; Postviral Syndrome; digital medicine
MeSH Terms: conditions — Inflammation; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This is a randomized two-arm, pre-post, clinical trial pilot study.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computerized Cognitive Remediation (Experimental)
  Interventions: Other: Computerized Cognitive Remediation
- Active Computer-Based Control (Active Comparator)
  Interventions: Other: Alternative Computer Activities

INTERVENTIONS:
Other: Computerized Cognitive Remediation — The computerized cognitive remediation intervention ("NeuroFlex") consists of a series of gamified tasks administered via computer tablet. The intervention provides both "bottom up" training to improve basic processing of sensory stimuli and "top down" training to improve executive functions. Importantly, NeuroFlex personalizes gameplay with adaptive algorithms that adjust difficulty on a trial-by-trial basis. Participants are prescribed a 30-hour dose distributed across 6 weeks. The treatment is completed remotely by the participant within their own home or other private location that is most convenient for the participant.
  Other Names: NeuroFlex
  Arms: Computerized Cognitive Remediation
Other: Alternative Computer Activities — The active control condition is carefully matched to the experimental condition in duration, computer tablet use, audiovisual stimulation, reward presentation, and interaction with study staff. It involves playing visuospatially-oriented computerized games that do not load on executive functions and watching stimulating educational videos.
  Arms: Active Computer-Based Control

SUMMARY:
The goal of this clinical trial is to determine if a neuroscience-based computerized cognitive remediation ("brain training") program can treat neurocognitive dysfunction (i.e., memory or thinking difficulties) that emerges in some older adults following a viral infection. The main questions it aims to answer are:

* Does computerized cognitive remediation improve cognitive performance and day-to-day functioning in older adults with postviral neurocognitive dysfunction?
* Will treatment effects be maintained over time, leading to better long term cognitive outcomes?
* Does the treatment lead to reductions in blood-based markers of inflammation as a potential mechanism of cognitive symptom improvement?
* Can the treatment be optimized and refined based on feedback from participants to improve user (patient) experience? Researchers will compare the computerized cognitive remediation program to an active computer-based control condition (alternative computer activities) to see if the computerized cognitive remediation program works to treat postviral neurocognitive dysfunction.

Participation takes approximately 43-48 hours over 7 months, with most activities (40-46 hours) completed within the first 7-8 weeks, including:

* Initial intake visit: Eligibility confirmation (~2-3 hours)
* Computer activities: About 5 hours per week for ~6 weeks (total ~30 hours) completed on a computer tablet provided by the study and loaned to participants for use during the treatment phase
* Weekly remote check-in meetings: ~30 minutes each during treatment
* Blood draws: Two sessions (before and after treatment), ~20-30 minutes each
* Three research visits: Pre-treatment, post-treatment, and 6-month follow-up (~2-3 hours each, including assessments of cognitive, emotional, and daily functioning)

DETAILED DESCRIPTION:
A significant minority of older adults display persistent cognitive impairments after the acute phase of a viral infection, referred to as Postviral Neurocognitive Dysfunction (PND). Underlying mechanisms remain poorly understood, though chronic neuroinflammation appears to reflect a key pathway. PND is debilitating, increases the risk for accelerated biological aging and dementia, and is associated with a substantial economic burden to society. Older adults are at heightened risk for PND given weakened immune systems, baseline age-related cognitive decline, and susceptibility to more severe acute viral illness. There is a critical lack of evidence-based treatments. The goal of this project is to determine the potential of a neuroplasticity-based computerized cognitive remediation (CCR) intervention for treating PND in older adults and probing underlying mechanisms.

The proposed design is a randomized, two-arm, clinical trial pilot study. Older adults with PND (N = 75) will be assigned to a 6-week course of neuroplasticity-based CCR or an active, computer-based control condition. Specific aims are to: examine preliminary efficacy of CCR for improving cognitive performance and day-to-day functioning in older adults with PND (Aim 1); optimize and refine the CCR program for older adults with PND using iterative, data-driven, participatory design methodology (Aim 2); and determine if CCR reduces peripheral inflammation as a potential mechanism of clinical symptom relief (Exploratory Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 60 years old
* prior history of COVID-19 that was confirmed with viral testing (e.g., positive laboratory test or positive at-home rapid test)
* cognitive symptoms (e.g., memory or thinking concerns) following COVID- 19 infection that have lasted for at least 12 weeks and are still present
* clinically meaningfully subjective cognitive concerns (i.e., T-score < 40) on the PROMIS-Cognitive Function Scale
* objective evidence of cognitive decline, as defined by performance on standardized measures of executive functioning, memory, or processing speed from the NIH Toolbox Cognition Battery that is at least 1 standard deviation below estimated premorbid cognitive functioning
* fluent in English language
* off psychiatric medication or on a stable dose for at least 8 weeks

Exclusion Criteria:

* history of neurological disorder with potential to interfere with study participation or confound results (e.g., uncontrolled seizure disorder, moderate to severe traumatic brain injury or stroke with persistent neurological deficits)
* history of dementia and/or dementia range performance on the Mini- Mental State Examination (i.e., score of less than or equal to 23)
* prior diagnosis of Mild Cognitive Impairment (MCI) or Mild Neurocognitive Disorder unrelated to the participant's history of COVID-19
* history of severe psychiatric illness that may interfere with study participation or confound results (e.g., bipolar disorder, schizophrenia, or other psychotic disorder)
* history of significant neurodevelopmental condition that may interfere with study participation or confound results (e.g., intellectual disability, autism spectrum disorder, or specific learning disorder with impairment in reading)
* alcohol or other substance use disorder within the past 2 years
* significant sensory impairments (e.g., blindness) that would interfere with the ability to complete neuropsychological measures or engage in the tablet-based intervention
* performance that is below expectation on a test of effort and validity

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-01-21 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Group Difference in Set-Shifting Abilities at Post-Treatment as Measured with Trails B | Pre-treatment and post-treatment (Week 7)
  Part B of the Trail Making Test (Trails B) is an executive functioning measure of set-shifting abilities in which the examinee must rapidly alternate between connecting numbers and letters distributed across a page. The total time (in seconds) required for the examinee to complete the task is recorded. Lower scores (in seconds) indicate better performance. Time to complete Trails B at the post-treatment visit will be compared between treatment groups (i.e., NeuroFlex vs. Active Control Condition), controlling for pre-treatment Trails B performance.
Group Difference in Set-Shifting Abilities at 6 Months as Measured with Trails B | Pre-treatment and 6 Months
  Part B of the Trail Making Test (Trails B) is an executive functioning measure of set-shifting abilities in which the examinee must rapidly alternate between connecting numbers and letters distributed across a page. The total time (in seconds) required for the examinee to complete the task is recorded. Lower scores (in seconds) indicate better performance. Time to complete Trails B at the 6-month visit will be compared between treatment groups (i.e., NeuroFlex vs. Active Control Condition), controlling for pre-treatment Trails B performance.
User Experience/Interface with Computerized Cognitive Remediation Program at Post-Treatment as Measured with the System Usability Scale | Post-Treatment (Week 7)
  The System Usability Scale is a well-validated, 10-item, self-report questionnaire of user experience/interface (UX/ UI) with computer-based programs. Participants rate each item using a 5-point Likert-style scale with response options ranging from "Strongly Disagree" to "Strongly Agree". Total scores ranging from 0-100 are calculated using a standard equation. Higher total scores indicate better UX/UI.

SECONDARY OUTCOMES:
Group Difference in Inhibitory Control at Post-Treatment as Measured with the Stroop Color and Word Test | Pre-treatment and post-treatment (Week 7)
  The Stroop Color and Word Test is an executive functioning measure of inhibitory control in which the examinee is presented with a sheet containing words of various colors printed in discordant ink colorings. The examinee is instructed to rapidly name the color of the ink that the words are printed in without reading the printed word (i.e., the prepotent response must be inhibited). An interference score is calculated by determining how many items the examinee completes within a set period of time, subtracting out their performance on baseline conditions (without an interference component) to control for processing speed. Higher scores indicate better performance. The score at the post-treatment visit will be compared between treatment groups (i.e., NeuroFlex vs. Active Control Condition), controlling for pre-treatment performance.
Group Difference in Inhibitory Control at 6 Months as Measured with the Stroop Color and Word Test | Pre-treatment and 6 months
  The Stroop Color and Word Test is an executive functioning measure of inhibitory control in which the examinee is presented with a sheet containing words of various colors printed in discordant ink colorings. The examinee is instructed to rapidly name the color of the ink that the words are printed in without reading the printed word (i.e., the prepotent response must be inhibited). An interference score is calculated by determining how many items the examinee completes within a set period of time, subtracting out their performance on baseline conditions (without an interference component) to control for processing speed. Higher scores indicate better performance. The score at the 6-Month visit will be compared between treatment groups (i.e., NeuroFlex vs. Active Control Condition), controlling for pre-treatment performance.
Group Difference in Verbal Generativity, Initiation, and Strategy Use at Post-Treatment as Measured with the Controlled Oral Word Association Test (COWAT) | Pre-treatment and post-treatment (Week 7)
  The COWAT is an executive functioning measure of verbal generativity, initiation, and strategy use in which the examinee must quickly generate as many words as possible, within a set period of time, according to pre-specified rules (e.g., words starting with a certain letter of the alphabet). A total score is calculated by adding up the number of words that were correctly produced within the time limit. Higher total scores indicate better performance. The score at the post-treatment visit will be compared between treatment groups (i.e., NeuroFlex vs. Active Control Condition), controlling for pre-treatment performance.
Group Difference in Verbal Generativity, Initiation, and Strategy Use at 6 Months as Measured with the Controlled Oral Word Association Test (COWAT) | Pre-treatment and 6-months
  The COWAT is an executive functioning measure of verbal generativity, initiation, and strategy use in which the examinee must quickly generate as many words as possible, within a set period of time, according to pre-specified rules (e.g., words starting with a certain letter of the alphabet). A total score is calculated by adding up the number of words that were correctly produced within the time limit. Higher total scores indicate better performance. The score at the 6-month visit will be compared between treatment groups (i.e., NeuroFlex vs. Active Control Condition), controlling for pre-treatment performance.
Group Difference in Attention-Related Problems at Post-Treatment as Measured with the Conners Continuous Performance Test | Pre-treatment and post-treatment (Week 7)
  The Conners Continuous Performance Test (Conners CPT) is a computerized measure of attention-related problems in which isolated letters are flashed briefly on a computer screen. The examinee is instructed to respond (by keypress) as quickly as possible whenever any letter appears on the screen, except for when the non-target letter appears. A summary measure of attention can be calculated based on the examinee's performance over the course of the test. The score at the post-treatment visit will be compared between treatment groups (i.e., NeuroFlex vs. Active Control Condition), controlling for pre-treatment performance.
Group Difference in Attention-Related Problems at 6 Months as Measured with the Conners Continuous Performance Test | Pre-treatment and 6-months
  The Conners Continuous Performance Test (Conners CPT) is a computerized measure of attention-related problems in which isolated letters are flashed briefly on a computer screen. The examinee is instructed to respond (by keypress) as quickly as possible whenever any letter appears on the screen, except for when the non-target letter appears. A summary measure of attention can be calculated based on the examinee's performance over the course of the test. The score at the 6-month visit will be compared between treatment groups (i.e., NeuroFlex vs. Active Control Condition), controlling for pre-treatment performance.
Group Difference in Subjective Cognitive Concerns at Post-Treatment as Measured with the Everyday Cognition Scale (ECog) | Pre-treatment and post-treatment (Week 7)
  The ECog is a self-report questionnaire of subjective cognitive concerns covering various domains, including memory, language, visuospatial skills, planning, organization, and divided attention. It uses a Likert-style scale ranging from 1-4, where 1 is "better or no change" and 4 is "consistently much worse" compared to prior. A total score, the average of all completed items ranging from 1 to 4, can be calculated to provide a global index of subjective cognitive concerns across domains. Lower total scores indicate better everyday cognitive functioning. The score at the post-treatment visit will be compared between treatment groups (i.e., NeuroFlex vs. Active Control Condition), controlling for pre-treatment performance.
Group Difference in Subjective Cognitive Concerns at 6 Months as Measured with the Everyday Cognition Scale (ECog) | Pre-treatment and 6-months
  The ECog is a self-report questionnaire of subjective cognitive concerns covering various domains, including memory, language, visuospatial skills, planning, organization, and divided attention. It uses a Likert-style scale ranging from 1-4, where 1 is "better or no change" and 4 is "consistently much worse" compared to prior. A total score, the average of all completed items ranging from 1 to 4, can be calculated to provide a global index of subjective cognitive concerns across domains. Lower total scores indicate better everyday cognitive functioning. The score at the 6-month visit will be compared between treatment groups (i.e., NeuroFlex vs. Active Control Condition), controlling for pre-treatment performance.
Group Difference in Functional Disability at Post-Treatment as Measured with the World Health Organization Disability Assessment Schedule (WHODAS) | Pre-treatment and post-treatment (Week 7)
  The WHODAS is a 36-item assessment instrument that measures functional disability in multiple domains, including cognition, mobility, selfcare, getting along (i.e., interacting with others), life activities, and participation (e.g., joining in community and societal activities). A summary score, ranging from 0 to 100, can be calculated that provides a measure of overall functioning across domains. Higher summary scores correspond to greater levels of functional disability. The score at the post-treatment visit will be compared between treatment groups (i.e., NeuroFlex vs. Active Control Condition), controlling for pre-treatment performance.
Group Difference in Functional Disability at 6 Months as Measured with the World Health Organization Disability Assessment Schedule (WHODAS) | Pre-treatment and 6-months
  The WHODAS is a 36-item assessment instrument that measures functional disability in multiple domains, including cognition, mobility, selfcare, getting along (i.e., interacting with others), life activities, and participation (e.g., joining in community and societal activities). A summary score, ranging from 0 to 100, can be calculated that provides a measure of overall functioning across domains. Higher summary scores correspond to greater levels of functional disability. The score at the 6-month visit will be compared between treatment groups (i.e., NeuroFlex vs. Active Control Condition), controlling for pre-treatment performance.
Group Difference in Episodic Memory at Post-Treatment as Measured with the California Verbal Learning Test (CVLT) | Pre-treatment and post-treatment (Week 7)
  The CVLT is a test of episodic memory that assesses the examinee's ability to learn and recall a list of words. The number of words correctly recalled after a delay period is measured (Long Delay Free Recall). Higher scores (i.e., more words recalled) correspond to better memory performance. The score at the post-treatment visit will be compared between treatment groups (i.e., NeuroFlex vs. Active Control Condition), controlling for pre-treatment performance.
Group Difference in Episodic Memory at 6 Months as Measured with the California Verbal Learning Test (CVLT) | Pre-treatment and 6-months
  The CVLT is a test of episodic memory that assesses the examinee's ability to learn and recall a list of words. The number of words correctly recalled after a delay period is measured (Long Delay Free Recall). Higher scores (i.e., more words recalled) correspond to better memory performance. The score at the 6-month visit will be compared between treatment groups (i.e., NeuroFlex vs. Active Control Condition), controlling for pre-treatment performance.

OTHER OUTCOMES:
Group Difference in Blood-Based Markers of Peripheral Inflammation at Post-Treatment | Pre-treatment and post-treatment (Week 7)
  Following manufacturer guidelines, concentrations of inflammatory markers (IL-6, TNF-alpha, and CRP) in plasma will be quantified using commercially available assays. Plasma concentrations at the post-treatment visit will be compared between treatment groups (i.e., NeuroFlex vs. Active Control Condition), controlling for pre-treatment concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Cutter Lindbergh, Ph.D., Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this project will be shared to enable analysis of the research findings described in the project aims. This includes individual subject level data on cognitive functioning, everyday functioning, cytokine concentrations, measures of intervention user experience, and pertinent demographics.
Supporting Information: Study Protocol
Time Frame: Data will be made available no later than the end of the performance period with no end date.
Access Criteria: It is planned to place anonymized data in a database called the National Archive of Computerized Data on Aging (NACDA). Access requires researchers to agree to refrain from sharing the data with others (no redistribution), not try to reidentify individuals, and to use the data only for research and statistical purposes. The information may be used for any type of research conducted in the future.
URL: https://www.icpsr.umich.edu/web/pages/NACDA/index.html